CLINICAL TRIAL: NCT00439244
Title: A One-year Partial Double-blinded, Randomized, Multi-center, Multi-national Study to Assess the Effects of Combination Therapy of Annual Zoledronic Acid (5 mg) and Daily Subcutaneous Teriparatide (2mcrg) on Postmenopausal Women With Severe Osteoporosis
Brief Title: Efficacy Study of Zoledronic Acid and Teriparatide Combination Therapy in Women With Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CZOL446H2409
Record Dates: First submitted 2007-02-22; First posted 2007-02-23 (Estimated); Results first posted 2011-04-20 (Estimated); Last update posted 2011-04-20 (Estimated); Status verified 2011-03

CONDITIONS: Osteoporosis
Keywords: Bone Mineral Density (BMD); C-Telopeptides (CTx); dual x-ray absorptiometry (DXA); pro-collagen type 1 N-propeptide (P1NP); teriparatide; zoledronic acid; Osteoporosis; postmenopausal women
MeSH Terms: conditions — Osteoporosis; Xanthomatosis, Cerebrotendinous | interventions — Zoledronic Acid; Teriparatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Zoledronic acid plus teriparatide (Active Comparator): Zoledronic acid 5.0 mg/100 mL was administered via a peripheral intravenous site at Visit 2 (once at randomization) as a slow 15-minute infusion. Teriparatide is supplied as sterile, colorless clear, isotonic solution in a glass cartridge which is pre-assembled into a disposable pen device for subcutaneous injection. The pen device delivers 20 μg of teriparatide concurrently as daily subcutaneous injections for 52 weeks.
  Interventions: Drug: Zoledronic acid; Drug: Teriparatide
- Zoledronic acid (Experimental): Zoledronic acid 5.0 mg/100 mL was administered via a peripheral intravenous site at Visit 2 (once at randomization) as a slow 15-minute infusion.
  Interventions: Drug: Zoledronic acid
- Placebo zoledronic acid plus teriparatide (Active Comparator): Placebo zoledronic acid 100 mL intravenous (i.v.) (once at randomization) plus teriparatide 20 μg (daily subcutaneous injections administered concurrently through 52 weeks). Teriparatide is supplied as sterile, colorless clear, isotonic solution in a glass cartridge which is pre-assembled into a disposable pen device for subcutaneous injection. The pen device delivers 20 μg of teriparatide concurrently as daily subcutaneous injections for 52 weeks.
  Interventions: Drug: Placebo; Drug: Teriparatide

INTERVENTIONS:
Drug: Zoledronic acid — Zoledronic acid 5.0 mg in a ready-to-infuse plastic bottle with a total fill volume of 103 mL to allow an infusion of 100 mL total volume corresponding to 5 mg of zoledronic acid.
  Other Names: Reclast, Aclasta
  Arms: Zoledronic acid; Zoledronic acid plus teriparatide
Drug: Placebo — Zoledronic acid matched placebo as a 103 mL solution of sterile water (physiologic 0.9% normal saline) to allow an infusion of 100 mL total volume in a ready-to-infuse plastic bottle
  Arms: Placebo zoledronic acid plus teriparatide
Drug: Teriparatide — Teriparatide is supplied as sterile, colorless clear, isotonic solution in a glass cartridge which is pre-assembled into a disposable pen device for subcutaneous injection. Each pre-filled delivery device is filled with 3.3 mL to deliver 3 mL.
  Each mL contains 250 μg teriparatide (corrected for acetate, chloride, and water content), 0.41 mg glacial acetate acid, 0.10 mg sodium acetate (anhydrous), 45.4 mg mannitol, 3.0 mg Metacresol, and water for injection. In addition, hydrochloric acid solution 10% and/or sodium hydroxide solution 10% may have been added to adjust the product to pH 4. Each cartridge pre-assembled into a pen device delivers 20 μg of teriparatide per dose each day for up to 28 days.
  Other Names: Forteo/Forsteo™
  Arms: Placebo zoledronic acid plus teriparatide; Zoledronic acid plus teriparatide

SUMMARY:
The purpose of this study is to assess the effects of zoledronic acid administered at the same time with teriparatide compared to zoledronic acid alone and teriparatide alone on bone mineral density (BMD) gain in the lumbar spine and total hip

ELIGIBILITY:
Inclusion criteria:

* Postmenopausal (PMO) women between 45 and 89 years of age.
* Bone mineral density T score of -2.5 or less at femoral neck, total hip or lumbar spine OR
* Bone mineral density T score of -2.0 or less at femoral neck, total hip or lumbar spine with at least one documented osteoporotic vertebral fracture or a previously documented history of an osteoporotic clinical non-vertebral fracture not due to excessive trauma

Exclusion criteria:

* Any prior use of strontium
* Any past or active kidney disease or problems with kidney function
* Prior treatment with any intravenous (i.v.) or oral bisphosphonate (such as but not limited to alendronate, risedronate and pamidronate) longer than 3 months consecutively. If bisphosphonate exposure is less than or equal to 3 months , a washout period of 1 year to randomization is required
* Calcium levels in blood within the normal range
* Normal liver function
* Non-osteoporotic forms of metabolic bone disease such as and not limited to Paget's disease of bone, osteomalacia, osteogenesis imperfecta or multiple myeloma
* Less than 3 evaluable lumbar (L1-L4) vertebrae for dual energy x-ray absorptiometry (DXA) measurement
* Treatment with osteoporotic therapies such as raloxifene, calcitonin or Hormone Replacement Therapy within 3 months of randomization
* Allergy or previous exposure to teriparatide

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 45 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2006-12; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (33):
- United States (18):
  - Birmingham, Alabama
  - Beverly Hills, California
  - Novartis Investigative Site, La Mesa, California
  - Novartis Investigative Site, Oakland, California
  - Colorado Springs, Colorado
  - Lakewood, Colorado
  - Gainesville, Georgia
  - Morton Grove, Illinois
  - Urbandale, Iowa
  - Bangor, Maine
  - Novartis Investigative Site, Woodbury, Minnesota
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Albuquerque, New Mexico
  - West Haverstraw, New York
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Spokane, Washington
  - Madison, Wisconsin
- Belgium (5):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative site, Godinne
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
- Germany (6):
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, München
  - Novartis Investigative site, Würzburg
- Spain (4):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Granada
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zoledronic Acid Plus Teriparatide | Zoledronic Acid | Placebo Zoledronic Acid Plus Teriparatide
Started | 137 ("Started" indicates randomized as well as intent to treat (ITT) population enrolled to study.) | 137 | 138
Safety Population | 137 (Total safety population is 411. One patient was randomized, but never received any study medication.) | 137 | 137
Completed | 126 | 131 | 131
Not Completed | 11 | 6 | 7
Not completed — Adverse Event | 5 | 2 | 3
Not completed — Withdrawal by Subject | 3 | 1 | 2
Not completed — Lost to Follow-up | 2 | 1 | 2
Not completed — Death | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Administrative problems | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoledronic Acid Plus Teriparatide | Zoledronic Acid | Placebo Zoledronic Acid Plus Teriparatide | Total
Number analyzed (Participants) | 137 | 137 | 138 | 412
Age Continuous [Mean (Standard Deviation); unit: years] | 65.0 (8.78) | 66.1 (9.02) | 63.8 (9.08) | 65.0 (8.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137 | 137 | 138 | 412
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Lumbar Spine Bone Mineral Density (BMD) at Week 52
Description: BMD measurements of the lumbar spine (L1-L4) by Dual X-ray absorptiometry (DXA) were performed on all patients at screening, and Weeks 13, 26, and 52 (or early termination). Every attempt was made to obtain the BMD measurements at the scheduled visit. If this was not possible, a BMD measurement ± 7 days from the scheduled visit was obtained. For the Final DXA at Week 52, the window was 10 - 15 days prior to the final study visit. BMD scans were acquired locally and all results sent to a central reader for evaluation.
Time Frame: Baseline through Week 52
Population: The intent-to-treat (ITT) population consisted of all randomized patients with available data.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Zoledronic Acid Plus Teriparatide | Zoledronic Acid | Placebo Zoledronic Acid Plus Teriparatide
Number analyzed (Participants) | 122 | 128 | 131
Percent change | 7.51 (0.414) | 4.37 (0.401) | 7.05 (0.398)

2. Secondary Outcome: Percent Change From Baseline in Lumbar Spine Bone Mineral Density (BMD) at Week 13 and Week 26
Description: as for outcome 1
Time Frame: Baseline through Week 13 and Week 26
Population: The intent-to-treat (ITT) population consisted of all randomized patients with available data. ITT patients with evaluable measurements at both baseline and post-baseline within each efficacy visit window were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Zoledronic Acid Plus Teriparatide | Zoledronic Acid | Placebo Zoledronic Acid Plus Teriparatide
Number analyzed (Participants) | 137 | 137 | 138
Percent Change
  At Week 13 (n= 127, 131, 131) | 4.65 (0.302) | 2.97 (0.297) | 2.88 (0.297)
  At Week 26 (n= 128, 130, 132) | 6.31 (0.337) | 3.87 (0.333) | 4.45 (0.330)

3. Secondary Outcome: Percent Change From Baseline in Total Hip Bone Mineral Density (BMD) at Week 13, Week 26 and Week 52
Description: BMD measurements of the total hip by Dual X-ray absorptiometry (DXA) were performed on all patients at screening, and Weeks 13, 26, and 52 (or early termination). Every attempt was made to obtain the BMD measurements at the scheduled visit. If this was not possible, a BMD measurement ± 7 days from the scheduled visit was obtained. For the final DXA at Week 52, the window was 10 - 15 days prior to the final study visit. BMD scans were acquired locally and all results sent to a central reader for evaluation.
Time Frame: Baseline through Week 13, Week 26 and Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Zoledronic Acid Plus Teriparatide | Zoledronic Acid | Placebo Zoledronic Acid Plus Teriparatide
Number analyzed (Participants) | 137 | 137 | 138
Percent Change
  At Week 13 (n= 127, 133, 133) | 2.54 (0.222) | 1.53 (0.216) | 0.75 (0.216)
  At Week 26 (n= 128, 130, 133) | 2.31 (0.265) | 1.73 (0.262) | 0.89 (0.259)
  At Week 52 (n= 123, 129, 129) | 2.33 (0.312) | 2.16 (0.303) | 1.10 (0.304)

4. Secondary Outcome: Bone Resorption and Formation Biochemical Markers : N-terminal Propeptide of Type I Collagen (P1NP)
Description: Specialized tests for markers of bone formation such as n-terminal propeptide of type I collagen (P1NP) were performed at Baseline, and Weeks 4, 8, 26, 39, and 52. The amount of serum P1NP was determined by the central laboratory.
Time Frame: At Baseline, Week 4, Week 8, Week 26, Week 39 and Week 52
Population: The intent-to-treat (ITT) population consisted of all randomized patients with available data. n = ITT patients with a measurement at each visit, as determined by the efficacy visit window
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Zoledronic Acid Plus Teriparatide | Zoledronic Acid | Placebo Zoledronic Acid Plus Teriparatide
Number analyzed (Participants) | 137 | 137 | 138
ng/mL
  At Baseline (n= 126, 129, 121) | 52.72 (24.815) | 53.64 (29.233) | 55.69 (28.631)
  At Week 4 (n= 109, 110, 104) | 61.74 (27.269) | 39.57 (20.532) | 93.63 (52.418)
  At Week 8 (n= 106, 107, 98) | 39.91 (22.412) | 21.68 (13.827) | 99.27 (48.404)
  At Week 26 (n= 116, 119, 114) | 65.26 (68.922) | 18.32 (15.255) | 156.97 (109.740)
  At Week 39 (n= 110, 115, 110) | 97.00 (112.804) | 20.69 (13.326) | 153.92 (103.065)
  At Week 52 (n= 110, 113, 112) | 112.87 (106.987) | 23.49 (16.137) | 137.53 (93.170)

5. Secondary Outcome: Bone Resorption and Formation Biochemical Markers : Beta C-terminal Telopeptides of Type I Collagen (β-CTx)
Description: Specialized tests for markers of bone formation such as β-CTx were performed at Baseline, and Weeks 4, 8, 26, 39, and 52. The amount of serum β-CTx was determined by the central laboratory.
Time Frame: At Baseline, Week 4, Week 8, Week 26, Week 39 and Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Zoledronic Acid Plus Teriparatide | Zoledronic Acid | Placebo Zoledronic Acid Plus Teriparatide
Number analyzed (Participants) | 137 | 137 | 138
ng/mL
  At Baseline (n= 126, 129, 121) | 0.45 (0.191) | 0.44 (0.218) | 0.46 (0.222)
  At Week 4 (n= 109, 110, 104) | 0.05 (0.048) | 0.05 (0.059) | 0.45 (0.259)
  At Week 8 (n= 106, 107, 98) | 0.09 (0.109) | 0.07 (0.112) | 0.60 (0.320)
  At Week 26 (n= 116, 119, 114) | 0.43 (0.419) | 0.12 (0.117) | 0.90 (0.537)
  At Week 39 (n= 110, 115, 110) | 0.57 (0.525) | 0.15 (0.108) | 0.89 (0.503)
  At Week 52 (n= 110, 113, 112) | 0.64 (0.476) | 0.17 (0.122) | 0.83 (0.393)

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: The safety population includes 411 patients, one less than the randomized population due to one patient who was randomized and never received any study medication.
Arm/Group | Zoledronic Acid | Zoledronic Acid Plus Teriparatide | Placebo Zoledronic Acid Plus Teriparatide
Serious Adverse Events (participants affected / at risk) | 20/137 | 13/137 | 15/137
Other Adverse Events (participants affected / at risk) | 115/137 | 118/137 | 96/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid (N=137) | Zoledronic Acid Plus Teriparatide (N=137) | Placebo Zoledronic Acid Plus Teriparatide (N=137)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 1
Right ventricular failure (Cardiac disorders) | 1 | 0 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 0 | 1
Glaucoma (Eye disorders) | 0 | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Face oedema (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0
Implant site irritation (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 1
Surgical failure (General disorders) | 0 | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
Stress urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0
Cystocele (Reproductive system and breast disorders) | 2 | 0 | 0
Rectocele (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Diaphragmatic hernia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Epiglottic cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Social problem (Social circumstances) | 0 | 1 | 0
Arterial haemorrhage (Vascular disorders) | 0 | 0 | 1
Arterial occlusive disease (Vascular disorders) | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 2 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid (N=137) | Zoledronic Acid Plus Teriparatide (N=137) | Placebo Zoledronic Acid Plus Teriparatide (N=137)
Vertigo (Ear and labyrinth disorders) | 7 | 5 | 9
Constipation (Gastrointestinal disorders) | 8 | 10 | 9
Diarrhoea (Gastrointestinal disorders) | 6 | 5 | 11
Dyspepsia (Gastrointestinal disorders) | 4 | 4 | 8
Nausea (Gastrointestinal disorders) | 15 | 21 | 19
Vomiting (Gastrointestinal disorders) | 9 | 10 | 4
Chills (General disorders) | 13 | 16 | 4
Fatigue (General disorders) | 17 | 19 | 13
Influenza like illness (General disorders) | 13 | 20 | 6
Oedema peripheral (General disorders) | 11 | 7 | 6
Pyrexia (General disorders) | 8 | 17 | 3
Bronchitis (Infections and infestations) | 17 | 5 | 6
Influenza (Infections and infestations) | 7 | 9 | 4
Nasopharyngitis (Infections and infestations) | 16 | 23 | 20
Sinusitis (Infections and infestations) | 5 | 7 | 1
Upper respiratory tract infection (Infections and infestations) | 7 | 5 | 7
Urinary tract infection (Infections and infestations) | 13 | 7 | 9
Contusion (Injury, poisoning and procedural complications) | 6 | 7 | 9
Fall (Injury, poisoning and procedural complications) | 9 | 7 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 | 31 | 18
Back pain (Musculoskeletal and connective tissue disorders) | 23 | 23 | 16
Bone pain (Musculoskeletal and connective tissue disorders) | 6 | 8 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 5 | 9
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 | 7 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 22 | 15 | 6
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 8 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 | 17 | 8
Dizziness (Nervous system disorders) | 3 | 5 | 7
Headache (Nervous system disorders) | 24 | 24 | 20
Hypertension (Vascular disorders) | 6 | 8 | 9

LIMITATIONS AND CAVEATS:
No teriparatide placebo available, Short study duration, Only bone mineral data, No bone strength or bone stucture assessment, No bone turnover markers data between 8 and 26 weeks, Study not powered for fracture outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.